CLINICAL TRIAL: NCT04810962
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of APP13007 for the Treatment of Inflammation and Pain After Cataract Surgery, Including a Corneal Endothelial Cell Sub-study
Brief Title: Efficacy and Safety of APP13007 for Treatment of Inflammation and Pain After Cataract Surgery Including a Corneal Endothelial Cell Sub-study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Formosa Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPN-302
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Ocular Inflammation and Pain After Cataract Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APP13007 0.05% BID (Experimental): 1 drop APP13007 0.05% twice daily for 14 days to study (operated) eye
  Interventions: Drug: APP13007, 0.05%
- Matching Vehicle Placebo (Placebo Comparator): 1 drop matching vehicle placebo twice daily for 14 days to study (operated) eye
  Interventions: Drug: Matching Vehicle Placebo for APP13007, 0.05%

INTERVENTIONS:
Drug: APP13007, 0.05% — APP13007 eye drop, 0.05%
  Arms: APP13007 0.05% BID
Drug: Matching Vehicle Placebo for APP13007, 0.05% — Matching vehicle placebo eye drop
  Arms: Matching Vehicle Placebo

SUMMARY:
This Phase 3 study will evaluate APP13007 in comparison to the matching vehicle placebo in a randomized, parallel-group, double-masked fashion. The subjects will have undergone routine cataract surgery on Day 0 of the study and will be assessed the next day (Post-operative Day; POD1) after uncomplicated surgery for eligibility for randomization to study treatment. The study comprises the Main Study and the Endothelial Cell Sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older expected to undergo unilateral uncomplicated cataract extraction via phacoemulsification and posterior chamber intraocular lens implantation in one eye.
* Have a pin-hole corrected visual acuity without other correction of ≤ 1.3 logarithm of the minimum angle of resolution (logMAR) in the study eye to be operated and contralateral eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart at Visit 1.
* Willing and able to comply with study requirements and visit schedule.
* Provide signed and dated informed consent.

Exclusion Criteria:

* Have a known sensitivity or allergy to clobetasol propionate, corticosteroids, or any of the study medication's components including benzalkonium chloride and soybean lecithin or any routine medication required during cataract surgery or for the conduct of study procedures
* Have an ACC count > 0 or any evidence of intraocular inflammation (e.g., flare) in either eye at the Screening visit
* Have a Grade > 0 on the Ocular Pain Assessment in either eye at the Screening visit

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — AimMax Therapeutics Inc.
Locations (31):
- United States (31):
  - Arizona Eye Center, Chandler, Arizona
  - Carrot Eye Center, Mesa, Arizona
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - Premiere Practice Management, LLC, Los Angeles, California
  - LoBue Laser and Eye Medical Center Inc, Murrieta, California
  - Visionary Research Institute, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Michael K. Tran, MD, Inc., Westminster, California
  - Rand Eye Institute, Deerfield Beach, Florida
  - Eye Associates for Fort Myers, Fort Myers, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - International Research Center, Tampa, Florida
  - Dixon Eye Care, Albany, Georgia
  - Clayton Eye Clinical Research LLC, Morrow, Georgia
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Stiles Eyecare Excellence and Glaucoma Institute, PA, Overland Park, Kansas
  - The Eye Care Center, Louisville, Kentucky
  - Fraser Eye Center, Fraser, Michigan
  - Ophthalmology Associates, St Louis, Missouri
  - Wellish Vision Institute, Las Vegas, Nevada
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - Alterman, Modi and Wolter, Poughkeepsie, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Eye Care Specialists, Kingston, Pennsylvania
  - Carolina Cataract and Laser Center, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Houston Eye Associates, Houston, Texas
  - DCT-Shah Research Institute LLC dba Discovery Clinical Trials, Mission, Texas
  - Round Rock Eye Consultants, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center US study in which 29 sites recruited subjects between March 2021 and March 2022.
Pre-assignment Details: Pre-assignment Details Of 466 enrolled participants, 370 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Started | 185 | 185
Completed | 179 | 179
Not Completed | 6 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — IP NOT AVAILABLE; REMAINED OUT OF THE COUNTRY; NON STUDY EYE NOT ELIGIBLE ON ENDOTHELIAL CELL COUNT | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo | Total
Number analyzed (Participants) | 185 | 185 | 370
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (9.7) | 68.0 (8.4) | 67.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 97 | 195
  Male | 87 | 88 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 35 | 73
  Not Hispanic or Latino | 147 | 150 | 297
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 17 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 20 | 22 | 42
  White | 150 | 145 | 295
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 185 | 185 | 370

OUTCOME MEASURES:

1. Primary Outcome: Participants With ACC Count = 0 in the Operated Study Eye at All Visits From Postoperative Day 8 Through Postoperative Day 15 Without Rescue Medication
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy at each study visit and the results are reported as number of cells in a 1mm x 1mm area.
Time Frame: Postoperative Day 8 and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 49 | 16
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

2. Primary Outcome: Participants With Ocular Pain Grade = 0 in the Operated Study Eye at All Visits From Postoperative Day 4 Through Postoperative Day 15 Without Rescue Medication
Description: Ocular pain is measured in the eye using a subject-reported five-point (0-4) ocular pain grade scale (0 = no pain; 1 = minimal; 2 = mild; 3 = moderate; 4 = severe pain).
Time Frame: Postoperative Day 4, Postoperative Day 8 and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 139 | 60
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

3. Primary Outcome: Participants With Treatment-emergent Adverse Events (AEs)
Description: Number of participants with ocular and systemic treatment-emergent AEs.
Time Frame: From First dose to Postoperative Day 22 (End of Main Study)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 184 | 185
Participants | 47 | 48

4. Secondary Outcome: Participants With Anterior Chamber Cell Grade = 0 in the Operated Study Eye at POD8 Without Rescue Medication
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy at each study visit and the results are reported as number of cells in a 1mm x 1mm area.ACC Grade 0 = 0 cells, ACC grade 1 = 1-5 cells, ACC grade 2 = 6-15 cells, ACC grade 3 = 16-30 cells, ACC grade 4 = >30 cells.
Time Frame: Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 55 | 24
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: Participants With Anterior Chamber Cell Grade = 0 in the Operated Study Eye at POD15 Without Rescue Medication
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy at each study visit and the results are reported as number of cells in a 1mm x 1mm area. ACC Grade 0 = 0 cells, ACC grade 1 = 1-5 cells, ACC grade 2 = 6-15 cells, ACC grade 3 = 16-30 cells, ACC grade 4 = >30 cells.
Time Frame: Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 107 | 35
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Participants With Ocular Pain Grade = 0 in the Operated Study Eye at POD4 Without Rescue Medication
Description: Ocular pain is measured in the eye using a subject-reported five-point (0-4) ocular pain grade scale (0 = no pain; 4 = severe pain).
Time Frame: Postoperative Day 4
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 158 | 95
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

7. Secondary Outcome: Participants With Ocular Pain Grade = 0 in the Operated Study Eye at POD8 Without Rescue Medication
Description: as for outcome 6
Time Frame: Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 161 | 86
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

8. Secondary Outcome: Participants With Ocular Pain Grade = 0 in the Operated Study Eye at POD15 Without Rescue Medication
Description: as for outcome 6
Time Frame: Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 160 | 92
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

9. Secondary Outcome: Participants With Anterior Chamber Flare (ACF) = 0 in the Operated Study Eye at POD4 Without Rescue Medication
Description: The degree of turbidity (flare) in the anterior chamber of the eye is measured using slit-lamp biomicroscopy and quantified on a five-point (0-4) anterior chamber flare grade scale (0 = none; 4 = Intense).
Time Frame: Postoperative Day 4
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 132 | 89
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

10. Secondary Outcome: Participants With Anterior Chamber Flare (ACF) = 0 in the Operated Study Eye at POD8 Without Rescue Medication
Description: as for outcome 9
Time Frame: Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 155 | 90
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

11. Secondary Outcome: Participants With Anterior Chamber Flare (ACF) = 0 in the Operated Study Eye at POD15 Without Rescue Medication
Description: as for outcome 9
Time Frame: Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 159 | 79
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

12. Secondary Outcome: Anterior Chamber Cell Grade in the Operated Study Eye - Change From Baseline (POD1 Prior to Dosing) to POD 15
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy and the results are reported as number of cells in a 1mm x 1mm area using a 5 point grading scale. ACC Grade 0 = 0 cells, ACC grade 1 = 1-5 cells, ACC grade 2 = 6-15 cells, ACC grade 3 = 16-30 cells, ACC grade 4 = >30 cells
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: grade on a scale
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
grade on a scale | -2.1 (0.1) | -1.0 (0.1)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -1.2, 95% CI 2-sided [-1.4 to -1.0] — Treatment Difference = APP13007-Placebo. Mean Difference Is the least-squares mean difference from the ANCOVA model with treatment as a fixed effect and baseline as a covariate

13. Secondary Outcome: Ocular Pain Grade in the Operated Study Eye - Change From Baseline (POD1 Prior to Dosing) to POD 15
Description: as for outcome 2
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: grade on a scale
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
grade on a scale | -0.6 (0.1) | -0.1 (0.1)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.7 to -0.3] — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Anterior Chamber Flare (ACF) in the Operated Study Eye - Change From Baseline (POD1 Prior to Dosing) to POD 15
Description: The degree of turbidity (flare) in the anterior chamber of the eye is measured using slit-lamp biomicroscopy and quantified on a five-point (0-4) anterior chamber flare grade scale (0 = none; 1 = faint; 2 = moderate; 3 = marked; 4 = Intense).
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: grade on a scale
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
grade on a scale | -0.6 (0.0) | -0.2 (0.0)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.5 to -0.3] — [estimate comment as in outcome 12, analysis 1]

15. Secondary Outcome: Best Corrected Visual Acuity in the Operated Study Eye - Change From Baseline (POD1 Prior to Dosing) to POD4
Description: The visual acuity in each eye is corrected using the pinhole method and the acuity is quantified on a logMAR (minimal angle of resolution) scale using the 'Early Treatment Diabetic Retinopathy Study' [ETDRS] charts for right and left eyes. A logMAR Score is calculated using the letter row on the chart and the number of incorrect letters read by the participant.
Time Frame: Baseline and Postoperative Day 4
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: logMAR Score
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
logMAR Score | -0.08 (0.01) | -0.03 (0.01)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.07 to -0.02] — [estimate comment as in outcome 12, analysis 1]

16. Secondary Outcome: Best Corrected Visual Acuity in the Operated Study Eye - Change From Baseline (POD1 Prior to Dosing) to POD8
Description: as for outcome 15
Time Frame: Baseline and Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: logMAR score
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
logMAR score | -0.11 (0.01) | -0.03 (0.01)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.10 to -0.05] — [estimate comment as in outcome 12, analysis 1]

17. Secondary Outcome: Best Corrected Visual Acuity in the Operated Study Eye - Change From Baseline (POD1 Prior to Dosing) to POD15
Description: as for outcome 15
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: logMAR score
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
logMAR score | -0.10 (0.01) | -0.02 (0.01)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.11 to -0.05] — [estimate comment as in outcome 12, analysis 1]

18. Secondary Outcome: Participants Using of Anti-inflammatory 'Rescue' Medication Through End-of-Treatment
Description: Participants who do not respond to study treatment after randomization are started on anti-inflammatory medication (referred to as 'Rescue' medication). The number of subjects starting 'Rescue' medication is recorded at each study visit
Time Frame: First dose to Postoperative Day 15
Population: Intent to Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 185 | 185
Participants | 13 | 71
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

19. Other Pre Specified Outcome: Corneal Endothelial Cell Density - Mean Change From Screening to Postoperative Day 85
Description: Corneal endothelial cell density in the Operated Study Eye (units: cells/mm2) was measured from the corneal endothelial cell images obtained using a specular microscope.
Time Frame: Screening and Postoperative Day 85
Population: Safety Population for Sub-study Participants
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 66 | 70
cells/mm2 | -276 (408) | -354 (437)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality data were collected from informed consent through Postoperative Day 85. Serious adverse events were collected from informed consent through Postoperative Day 85. Other (not Including Serious) adverse events were collected from the first dose through Postoperative Day 22 (end of Main Study).
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/185
Serious Adverse Events (participants affected / at risk) | 1/184 | 4/185
Other Adverse Events (participants affected / at risk) | 6/184 | 14/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APP13007 0.05% BID (N=184) | Matching Vehicle Placebo (N=185)
Cystoid macular oedema (Eye disorders) | 1 (1) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APP13007 0.05% BID (N=184) | Matching Vehicle Placebo (N=185)
Eye inflammation (Eye disorders) | 6 (6) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institutions and Investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT04810962/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT04810962/SAP_001.pdf